CLINICAL TRIAL: NCT07006792
Title: A Phase 4, Multicenter, Open-label, Single-arm Study to Investigate the Efficacy of Lebrikizumab in Adult and Adolescent Participants With Moderate Atopic Dermatitis and High Itch Burden
Brief Title: A Study to See How Well Lebrikizumab Works in Adults and Adolescents With Moderate Atopic Dermatitis (Eczema) and High Itch Burden
Acronym: ADsolve
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27407; J2T-MC-KGCE (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — lebrikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lebrikizumab (Experimental): Lebrikizumab administered subcutaneously (SC).
  Interventions: Drug: Lebrikizumab

INTERVENTIONS:
Drug: Lebrikizumab — Administered SC
  Other Names: LY3650150

SUMMARY:
The purpose of this study is to measure how well taking lebrikizumab alone works for participants with fewer places on the body with eczema (atopic dermatitis), but these places may be very itchy.

Participation in this study will last up to approximately 38 weeks (9 and a half months) including 24 weeks (6 months) of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic atopic dermatitis (AD) (according to American Academy of Dermatology Consensus Criteria) that has been present for ≥1 year before screening visit.
* Have 10% to 25% body surface area (BSA) of AD involvement at screening and baseline.
* Have pruritus numeric rating scale (NRS) ≥6 at baseline.
* Have an Eczema Area and Severity Index (EASI) score ≥16 at screening and baseline.
* Have an Investigator's Global Assessment (IGA) score ≥3 (on a scale of 0 to 4) at screening and baseline.
* Based on investigator judgement, have a history of inadequate response to treatment with topical medications, or determination that topical treatments are otherwise medically inadvisable.
* For participants aged 12 to less than 18, have a body weight ≥40 kilograms (kg) at baseline.

Exclusion Criteria:

* Have an uncontrolled chronic disease that might require multiple intermittent uses of oral corticosteroids at screening (as defined by the investigator).
* Have known liver cirrhosis and/or chronic hepatitis of any etiology.
* History of malignancy, including mycosis fungoides or cutaneous T-cell lymphoma, within 5 years before the screening, except completely treated in situ carcinoma of the cervix of completely treated and resolved nonmetastatic squamous or basal cell carcinoma of the skin with no evidence of recurrence in the past 12 weeks.
* Are diagnosed with active endoparasitic infections or at high risk of these infections.
* Have a known or suspected history of immunosuppression, including history of invasive opportunistic infections despite infection resolution; or unusually frequent, recurrent, or prolonged infections, per the investigator's judgment.
* Have presence of skin comorbidities that may interfere with study assessments.
* Have a severe concomitant illness(es) that in the investigator's judgment would adversely affect the participant's participation in the study.
* Have had any of the following types of infection within 3 months of screening or develop any of these infections during screening:

  * Serious (requiring hospitalization, and/or intravenous or equivalent oral antibiotic treatment).
  * Opportunistic - Note: Herpes zoster is considered active and ongoing until all vesicles are dry and crusted over.
  * Chronic (duration of symptoms, signs, and/or treatment of 6 weeks or longer).
  * Recurring (including, but not limited to, recurring cellulitis and chronic osteomyelitis).
* Have an active or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before the baseline visit or superficial skin infections within 1 week before the baseline visit.
* Have had any prior treatment with a biologic therapy for AD.
* Have had treatment with any of the following agents within 4 weeks prior to the baseline visit:

  * systemic immunosuppressive or immunomodulating drugs (for example, systemic corticosteroids, cyclosporine, mycophenolate mofetil, interferon-gamma,
  * azathioprine, methotrexate, and other immunosuppressants)
  * small molecules (for example, Janus kinase inhibitors [topical or systemic]), or
  * phototherapy and photochemotherapy for AD.
* Treatment with B-cell-depleting biologics, including rituximab, within 6 months prior to baseline.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Eczema Area and Severity Index-75 (EASI-75) (≥75% Reduction from Baseline in EASI), or a ≥4-point Reduction in Pruritus Numerical Rating Scale (NRS) from Baseline | Week 16
  The primary endpoint will be a composite endpoint as defined by achieving either EASI-75 or Pruritus NRS≥4-point Reduction from Baseline.

SECONDARY OUTCOMES:
Percentage of Participants Achieving EASI-75 | Baseline to Week 24
Percentage of Participants Achieving a ≥4-point Reduction from Baseline in Pruritus NRS | Baseline to Week 24
Percentage of Participants with an Investigator's Global Assessment (IGA) of 0 or 1 and a Reduction ≥2 points from Baseline | Baseline to Week 24
Percentage of Participants Achieving EASI-90 | Baseline to Week 24
Change from Baseline in Body Surface Area (BSA) Involvement | Baseline, Week 24
Percentage of Change from Baseline in Pruritus NRS Score | Baseline, Week 24
Percentage of Participants with a Sleep-loss Scale Score of ≥2 points at Baseline Who Achieve a ≥ 2-point Reduction | Baseline to Week 24
Percentage Change from Baseline in Sleep-loss Scale | Baseline, Week 24
Percentage of Participants with a Skin Pain NRS of ≥4 Points at Baseline Who Achieve a ≥4-point Reduction | Baseline to Week 24
Change from Baseline in Dermatology Quality of Life (DLQI) | Baseline, Week 24
Change from Baseline in Children's Dermatology Quality of Life (CDLQI) | Baseline, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (73):
- United States (39):
  - Total Skin & Beauty Dermatology Center, PC DBA Total Dermatology, Birmingham, Alabama
  - Research Solutions of Arizona, Litchfield Park, Arizona
  - Alliance Dermatology and Mohs Center, Phoenix, Arizona
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - First OC Dermatology Research Inc, Fountain Valley, California
  - Dermatology Research Associates, Los Angeles, California
  - NorCal Clinical Research, Rocklin, California
  - Suncoast Research Associates, Doral, Florida
  - Encore Medical Research, Hollywood, Florida
  - Solutions Through Advanced Research, Jacksonville, Florida
  - Life Arc Research Centers - Miami, Miami, Florida
  - MCR Research, Miami, Florida
  - Health Clinical Research, Miami, Florida
  - Deluxe Health Center, Miami Lakes, Florida
  - Renstar Medical Research, Ocala, Florida
  - Leading Edge Dermatology, Plantation, Florida
  - Research Institute of the Southeast, West Palm Beach, Florida
  - Dermatology Affiliates Research Institute, Atlanta, Georgia
  - DeNova Research, Chicago, Illinois
  - Southern Indiana Clinical Research Center, Columbus, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Southern Indiana Clinical Trials, New Albany, Indiana
  - Equity Medical - Bowling Green, Bowling Green, Kentucky
  - Allergy & Asthma Specialists, P.S.C., Owensboro, Kentucky
  - Foxhall Research Center, Chevy Chase, Maryland
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Revival Research Institute, LLC, Troy, Michigan
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Equity Medical, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Hickory Dermatology Research Center, Hickory, North Carolina
  - Dermatologists of Central States, LLC, Fairborn, Ohio
  - ObjectiveHealth - Goodlettsville Dermatology Research, Goodlettsville, Tennessee
  - John Peter Smith Hospital, Fort Worth, Texas
  - Reveal Research Institute - Frisco, Frisco, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Prime Clinical Research - Mansfield, Mansfield, Texas
  - Texas Dermatology and Laser Specialists - San Antonio - South New Braunfels Avenue, San Antonio, Texas
  - Jordan Valley Dermatology & Research Center, South Jordan, Utah
- Argentina (11):
  - CONEXA Investigacion Clinica S.A., Buenos Aires
  - CIPREC, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - DOM Centro de Reumatología, Buenos Aires
  - Instituto de Neumonologia Y Dermatologia, Buenos Aires
  - Psoriahue, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Parra Dermatología, Mendoza
  - INECO Neurociencias Oroño, Rosario
  - Instituto de Investigaciones Clinicas Rosario, Rosario
  - Centro de Investigaciones San Miguel, San Miguel
- Brazil (9):
  - AlergoAlpha - Barueri, Barueri
  - PUC Trials- Nucleo de Pesquisa clinica da Escola de Medicina da PUCPR, Curitiba
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Hospital São Lucas da PUCRS, Porto Alegre
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - Centro de Pesquisas da Clínica IBIS, Salvador
  - Faculdade de Medicina do ABC, Santo André
  - ISPEM - Instituto São José dos Campos em Pesquisas Médicas, São José dos Campos
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
- Canada (12):
  - Dermatology Research Institute, Calgary
  - Skin Physicians Dermatology, Edmonton
  - Brunswick Dermatology Center, Fredericton
  - Maritime Dermatology, Halifax
  - Lovegrove Dermatology, London
  - Skin Care West, Nanaimo
  - Kanata Allergy Clinic, Ottawa
  - SKiN Centre for Dermatology, Peterborough
  - Oak Ridges Aesthetics Centre, Richmond Hill
  - Centre de Recherche Saint-Louis, Sherbrooke
  - Eternal Springtime Dermatology, Thunder Bay
  - North York Research Inc, Toronto
- Puerto Rico (2):
  - Dr. Samuel Sanchez PSC, Caguas
  - CMRC Headlands, LLC, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/